CLINICAL TRIAL: NCT06213259
Title: A Phase 1, Randomised, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Pharmacodynamics of KD6005 in Healthy Participants and Participants With Rheumatoid Arthritis (RA).
Brief Title: A Study of KD6005 in Healthy Participants and Participants With Rheumatoid Arthritis (RA)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Kanda Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KD6005CT01
Record Dates: First submitted 2023-12-25; First posted 2024-01-19 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2023-12

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- KD6005 (Healthy) (Experimental): Healthy participants will receive a single dose of KD6005 in dose escalation cohorts subcutaneously (SQ).
  Interventions: Drug: KD6005
- Placebo (Healthy) (Placebo Comparator): Healthy participants will receive a single dose of placebo, SQ.
  Interventions: Drug: Placebo
- KD6005(RA) (Experimental): Participants with RA will receive a multiple-dose of KD6005 in dose escalation cohorts, SQ.
  Interventions: Drug: KD6005
- Placebo (RA) (Placebo Comparator): Participants with RA will receive a multiple-dose of placebo, SQ.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KD6005 — Biological: KD6005, SQ
  Arms: KD6005 (Healthy); KD6005(RA)
Drug: Placebo — Placebo, SQ
  Arms: Placebo (Healthy); Placebo (RA)

SUMMARY:
This phase 1 study will consist of two parts: Phase 1a is a single-dose study, and will evaluate the safety, tolerability, pharmacokinetics (PK) and preliminary pharmacodynamics (PD) in healthy participants. Phase 1b is a multiple doses study, and will evaluate the safety, tolerability, PK and preliminary PD in participants with rheumatoid arthritis (RA).

ELIGIBILITY:
Inclusion Criteria:

Main Inclusion Criteria for Healthy Participants (Phase 1a):

1. Being voluntary to sign the informed consent form.
2. Male or female age 18 to 50 years. Have a body mass index (BMI) between 19 and 26 kg/m2 inclusive and weigh at least 50kg for male , or at least 45kg female. In good overall health at the time of screening.

Main Inclusion Criteria for RA participants (Phase 1b):

1. Being voluntary to sign the informed consent form.
2. Age 18-70 years old, and subjects with rheumatoid arthritis (RA) diagnosed by the 1987 or 2010 American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) classification criteria.

Exclusion Criteria:

Main Exclusion Criteria for Healthy Participants (Phase 1a):

1. Known to be allergic to KD6005 or its components.
2. History of malignancy under study within 5 years, except adequately treated and cured basal or squamous cell carcinoma of the skin or cervical carcinoma in situ.
3. Subjects who had undergone any surgical procedures within 3 months prior to screening, or will plan surgery during the study period and within 1 month after the study ended.
4. History of clinically significant cardiovascular, hepatic, neurological, respiratory, hematological, digestive, rheumatological, immune, renal, or psychiatric disorders that the investigator believes may confuse the study results or place the subject at undue risk.
5. Subjects who are judged by the investigator to have a disease affecting drug absorption, distribution, metabolism, and excretion; Or skin disease or other disease affecting subcutaneous injection.
6. Clinical symptoms, signs, laboratory tests or X-ray tests suggest active tuberculosis(TB).
7. An infection that the investigators determined to be clinically significant occurred within 3 months prior to screening.
8. Blood donation within the last 3 months (more than 400mL).
9. Subjects who have participated in clinical trials of any drug or medical device within 3 months or 5 drug half-lives (whichever is longer) prior to screening.
10. Any acute illness that the investigators determined to be clinically significant occurred in the 1 month prior to screening.
11. A history of severe herpes virus infection.
12. A history of drug use or substance abuse.
13. Subjects who received live/attenuated vaccine within 2 months prior to screening or required live vaccines during study participation, including within 28 days after the last KD6005 administration.
14. Received any medication within 4 weeks prior to use of KD6005.
15. Subjects who have been tested positive for the following tests: Hepatitis B virus (HBV), Hepatitis C virus (HCV), human immunodeficiency virus (HIV).
16. Pregnant or breastfeeding females.
17. Smoke greater than 5 cigarettes/day.
18. Alcoholism: Positive breath test for alcohol.
19. Subjects who may not be able to complete the study for other reasons or who the investigator believes should not be included.

Main Exclusion Criteria for RA participants (Phase 1b):

1. History of congestive heart failure, including asymptomatic congestive heart failure.
2. History of serious diseases of hepatic, renal and other important organs, hematological and endocrine system disorders.
3. Subjects diagnosed with other rheumatic immune system diseases, except rheumatoid arthritis secondary sjogren's syndrome and asymptomatic Hashimoto thyroiditis.
4. Severe infection or acute or chronic infection in the 6 months prior to the initial study.
5. History of latent or active granulomatous infection in the 6 months prior to screening.
6. History of a non-tuberculous mycobacterium infection or an opportunistic infection within 6 months prior to screening.
7. Present or previous history of malignant tumor.
8. Pregnant or breastfeeding females.
9. Subjects who have participated in clinical trials of any drug within 3 months prior to screening.
10. Subjects who received live vaccine within 3 months prior to screening, or who will plan to receive live vaccine within 3 months from the first administration to the last administration of the KD6005.
11. Treatment with small-molecule targeted drugs, such as JAK inhibitors, within 4 weeks prior to randomization.
12. HBV screening includes HbsAg (surface antigen), anti-HBs (surface antibody) and anti-HBc (core antibody). Evidence of hepatitis B infection (positive for HBsAg).
13. Subjects with a positive test for tuberculosis (TB).
14. Subjects who have been tested positive for the following tests: Hepatitis C virus (HCV), human immunodeficiency virus (HIV).
15. Known to be allergic to the KD6005.
16. Subjects with a joint functional class IV or those who are bedridden or wheelchair-bound for a long time.
17. Subjects with arthritic diseases other than osteoarthritis.
18. Subjects have depression or the significant suicide ideation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-01-06 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Phase 1a, and Phase 1b: The incidence and safety profile of participants with adverse events (AEs), serious adverse events(SAE) | Phase 1a: Through study completion, an average of 42 Days; Phase 1b: Through study completion, an average of 57 Days
  To assess the safety and tolerability of KD6005 in healthy participants or Rheumatoid Arthritis (RA) participants.
Phase 1a, and Phase 1b: Percentage of Participants With Laboratory Abnormalities, that have clinical significance | Phase 1a: Through study completion, an average of 42 Days; Phase 1b: Through study completion, an average of 57 Days
Phase 1a: The Pharmacokinetics(PK) profile of KD6005: Maximum observed serum concentration (Cmax) | Through study completion, an average of 42 Days
Phase 1a: The Pharmacokinetics(PK) profile of KD6005: Time to reach maximum serum concentration (Tmax) | Through study completion, an average of 42 Days
Phase 1a: The Pharmacokinetics(PK) profile of KD6005: half-life (T1/2) | Through study completion, an average of 42 Days
Phase 1a: The Pharmacokinetics(PK) profile of KD6005: Area under blood concentration-time curve (AUC0-T and AUC0-∞) | Through study completion, an average of 42 Days
Phase 1a: The Pharmacokinetics(PK) profile of KD6005: Apparent volume of distribution (Vd) | Through study completion, an average of 42 Days
Phase 1a: The Pharmacokinetics(PK) profile of KD6005: Mean retention time (MRT) | Through study completion, an average of 42 Days

SECONDARY OUTCOMES:
Phase 1a, and Phase 1b: The immunogenicity of KD6005 | Phase 1a: Through study completion, an average of 42 Days; Phase 1b: Through study completion, an average of 57 Days
  Including the incidence of ADA positive. For ADA positive patients, the incidence of neutralizing antibody (NAB) will be analyzed.
Phase 1b: The Pharmacokinetics(PK) profile of KD6005: Maximum observed serum concentration (Cmax) | Through study completion, an average of 57 Days
Phase 1b: The Pharmacokinetics(PK) profile of KD6005: Time to reach maximum serum concentration (Tmax) | Through study completion, an average of 57 Days
Phase 1b: The Pharmacokinetics(PK) profile of KD6005: half-life (T1/2) | Through study completion, an average of 57 Days
Phase 1b: The Pharmacokinetics(PK) profile of KD6005: Area under blood concentration-time curve (AUC0-T and AUC0-∞) | Through study completion, an average of 57 Days
Phase 1b: The Pharmacokinetics(PK) profile of KD6005: Apparent volume of distribution (Vd) | Through study completion, an average of 57 Days
Phase 1b: The Pharmacokinetics(PK) profile of KD6005: Mean retention time (MRT) | Through study completion, an average of 57 Days
Phase 1b: Change From Baseline in Erythrocyte sedimentation rate (ESR) | Through study completion, an average of 57 Days
  Preliminary pharmacodynamic evaluation in RA participants.
Phase 1b: Change From Baseline in C-reactive protein (CRP) | Through study completion, an average of 57 Days
  Preliminary pharmacodynamic evaluation in RA participants.
Phase 1b: Change From Baseline in anti-Cyclic citrullinated peptide antibody (anti-CCP) | Through study completion, an average of 57 Days
  Preliminary pharmacodynamic evaluation in RA participants.
Phase 1b: Percentage of Participants Who Achieved an American College of Rheumatology (ACR) 20% Improvement (ACR20) Response | Through study completion, an average of 57 Days
  Preliminary pharmacodynamic evaluation in RA participants.
Phase 1b: Percentage of Participants Who Achieved an American College of Rheumatology (ACR) 50% Improvement (ACR50) Response | Through study completion, an average of 57 Days
  Preliminary pharmacodynamic evaluation in RA participants.
Phase 1b: Percentage of Participants Who Achieved an American College of Rheumatology (ACR) 70% Improvement (ACR70) Response | Through study completion, an average of 57 Days
  Preliminary pharmacodynamic evaluation in RA participants.
Phase 1b: Change From Baseline in Disease Activity Score for 28 Joint Counts (DAS28) Using CRP | Through study completion, an average of 57 Days
  Preliminary pharmacodynamic evaluation in RA participants.
Phase 1b: Change From Baseline in Disease Activity Score for 28 Joint Counts (DAS28) Using ESR | Through study completion, an average of 57 Days
  Preliminary pharmacodynamic evaluation in RA participants.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Fang, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, China